CLINICAL TRIAL: NCT02650479
Title: Two-Part, Randomized, Placebo and Active-Controlled, Double-Blind, Thorough QT Study Evaluating the Effects of Intravenous Exenatide on Cardiac Repolarization in Healthy Male and Female Volunteers
Brief Title: Study of the Effects of Intravenous Exenatide on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITCA-650-CLP-114
Record Dates: First submitted 2016-01-01; First posted 2016-01-08 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Adult Male and Female Volunteers
MeSH Terms: interventions — Exenatide; Moxifloxacin; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IV exenatide - pilot study (Other): IV Exenatide Infusion 0.1250 mcg/kg/hour for 0.5 hours followed by 0.0625 mcg/kg/hour for 5.5 hours, preceded by IV Palonosetron 0.25 mg for nausea/vomiting prophylaxis.
  Interventions: Drug: Exenatide; Drug: Palonosetron
- Treatment Group A - core study (Experimental): IV Exenatide Infusion 0.1250 mcg/kg/hour for 0.5 hours followed by 0.0625 mcg/kg/hour for 5.5 hours, preceded by IV Palonosetron 0.25 mg for nausea/vomiting prophylaxis.
  Interventions: Drug: Exenatide; Drug: Palonosetron
- Treatment Group B - core study (Experimental): IV infusion of placebo over 6 hours, preceded by IV Palonosetron 0.25 mg for nausea/vomiting prophylaxis.
  Interventions: Drug: Placebo; Drug: Palonosetron
- Treatment Group C - core study (Experimental): IV infusion of placebo over 6 hours and a single oral dose of 400 mg moxifloxacin within 1 min of start of infusion, preceded by IV Palonosetron 0.25 mg for nausea/vomiting prophylaxis.
  Interventions: Drug: Placebo; Drug: Moxifloxacin; Drug: Palonosetron

INTERVENTIONS:
Drug: Exenatide — 6 hour IV infusion (double infusion of 0.1250 mcg/kg/hour for 30 min followed by infusion rate (1X) of 0.0625 mcg/kg/hour for 5.5 hours).
  Arms: IV exenatide - pilot study; Treatment Group A - core study
Drug: Placebo — 6 hour IV infusion.
  Arms: Treatment Group B - core study; Treatment Group C - core study
Drug: Moxifloxacin — 400 mg oral dose moxifloxacin within 1 min of start of infusion of exenatide
  Arms: Treatment Group C - core study
Drug: Palonosetron — 0.25 mg administered IV within 30 minutes prior to initiating the infusion of exenatide

SUMMARY:
Two-Part, Randomized, Placebo and Active-Controlled, Double-Blind, Thorough QT Study Evaluating the Effects of Intravenous Exenatide on Cardiac Repolarization in Healthy Male and Female Volunteers

DETAILED DESCRIPTION:
This single-center Phase I study will consist of 2 parts, a Pilot Part and a Core Part.

The Pilot Part of the study will be an open-label, non-randomized, single-treatment design in 10 healthy male and female subjects to determine if an infusion regimen of a 6-h continuous IV infusion of exenatide will lead to a mean plasma steady state concentration of 500 pg/mL.

The Core part of the study will be a double-blind (except for the use of open label active control moxifloxacin), randomized, placebo-controlled,3 period, 6-sequence, cross-over design in 72 healthy male and female subjects to evaluate whether exenatide at therapeutic and supra-therapeutic concentrations has a pharmacological effect on cardiac repolarization (threshold value >10 msec).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 19 to 35 kg/m2 inclusive.
* Women of child bearing potential - use of an additional adequate method of contraception during the study and until 1 additional menstrual cycle following the end-of-study (EOS) visit. Adequate methods of contraception for women of child bearing potential (WOCBP) include: mechanical products (ie, intrauterine device [IUD]-copper IUD); or barrier methods (eg, diaphragm, condoms, cervical cap) with spermacide.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), and bilirubin within normal range at Screening.
* Fasting triglycerides within the normal range at Screening

Exclusion Criteria:

* History of type 1 or type 2 diabetes, or history of hypoglycemia.
* History or evidence of myocardial infarction, congestive heart failure, syncope not related to heart arrhythmia, coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention), unstable angina, or cerebrovascular accident or stroke or TIA.
* History of atrial fibrillation, flutter, or non-sustained or sustained VT.
* Personal or family history of sudden death or long QT syndrome.
* History of uncontrolled hypertension.
* History or evidence of acute or chronic pancreatitis.
* History of liver disease.
* Abnormal renal function.
* History of medullary thyroid cancer or a personal or family history of multiple endocrine neoplasia type 2.
* Thyroid-stimulating hormone (TSH) outside of normal limits at Screening .
* Weight loss surgery.
* History of malignancy (not including basal or squamous cell carcinoma of the skin with past 5 years). (Subjects who have been disease free for greater than 5 years may be included.)
* History of active alcohol within 1 year prior to Screening.
* History of drug abuse within 5 years prior to Screening or a positive prestudy drug screen.
* Weekly consumption of more than 14 alcoholic beverages for females and more than 21 alcoholic beverages for males.
* Smoke more than 10 cigarettes per day.
* Excessive in xanthine consumption (more than 5 cups of coffee or equivalent per day).
* History of hypersensitivity to any of the medications used in this study.
* Women that are pregnant, lactating, or planning to become pregnant.
* History of or positive results on screening tests for hepatitis B and/or hepatitis C and/or human immunodeficiency virus (HIV).
* History or evidence of immunocompromised status.
* Prior or current treatment with any GLP-1 receptor agonist (eg, Bydureon™, Byetta®, Victoza®, Tanzeum® or exogenous native GLP-1) or prior participation in an ITCA 650 clinical trial.
* Any gastrointestinal complaints within 7 days prior to first dosing.
* Use of medications within 14 days of first dose other than hormone replacement therapy and oral contraceptives.
* Chronic (8 consecutive days or greater) treatment with systemic corticosteroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pilot Study: Establishment of mean plasma steady state concentration of 500 pg/mL | 35 days
Core Study: Changes to QTc interval changes (threshold > 10 msec) measurements | 56 days

SECONDARY OUTCOMES:
Pilot Study: Adverse events as assessed by subjective subject reporting, laboratory testing, ECG, physical examinations, and vital signs | 35 days
Core Study: Measurement of exenatide plasma concentrations and relationship to changes in QTc interval measurements | 56 days
  Relationship between plasma concentrations of exenatide and QTc interval.
Core Study: Changes in PR, RR, QRS, QT, T- and U- wave morphology | 56 days
Core Study: Measurement of QTc interval changes moxifloxacin as active control | 56 days
Core Study: Adverse events as assessed by subjective subject reporting, laboratory testing, ECG, physical examinations, and vital signs | 56 days
Pilot Study: Maximum concentration (CMax) of exenatide | 35 days
Pilot Study: Time to maximum concentration (TMax) of exenatide | 35 days
Pilot Study: Area under the curve (AUC) of exenatide | 35 days
Pilot Study: Steady state concentration (Css) of exenatide | 35 days
Pilot Study: Half life (T1/2) of exenatide | 35 days
Core Study: Half life (T1/2) of exenatide | 56 days
Core Study: Steady state concentration (Css) of exenatide | 56 days
Core Study: Area under the curve (AUC) of exenatide | 56 days
Core Study: Maximum concentration (CMax) | 56 days
Core Study: Time to maximum concentration (TMax) of exenatide | 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- PRA-Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No